CLINICAL TRIAL: NCT06565767
Title: Continuous Chest Compressions Training Among Schoolchildren With Gamification in Brazil: a Pilot Study Study Start Date November 2022
Brief Title: Continuous Chest Compressions Training Among Schoolchildren With Gamification in Brazil: a Pilot Study
Acronym: CSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: University of Marília (Unknown); INVITARE Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 161976
Record Dates: First submitted 2024-08-06; First posted 2024-08-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Cardiopulmonary Resuscitation; Educational Problems

STUDY DESIGN:
Masking Description: open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): age 7 to 11
  Interventions: Other: cardiopulmonary resuscitation quality
- Group 2 (Experimental): age 11 to 17
  Interventions: Other: cardiopulmonary resuscitation quality

INTERVENTIONS:
Other: cardiopulmonary resuscitation quality — variability in compression depth among different age groups, taking into account physical attributes, through an active learning approach and game-based learning framework

SUMMARY:
This study employed a randomized cluster intervention design to evaluate differences in chest compression depth among children's groups, using active learning methodologies and serious game-based learning as part of the Kids Save Hearts Project.

DETAILED DESCRIPTION:
A cluster randomized trial will be carried out where the distribution among groups will be conducted by block. Four hundred children from elementary and high school will be included, divided into two groups based on age: 7 to 10 years (Group I) and 11 to 17 years (Group II). The selection of groups will be performed through randomization using the Research Randomizer computer software (www.randomizer.org) among 20 schools (public and private) of the state of São Paulo, Brazil. An appropriate number of classes will be enrolled to match the sample size, considering a mean value of 20 students per class. The study will be conducted from 2022 to 2026. Schoolchildren and their legal guardians will give written informed assent and consent to participate in the study. The inclusion criteria will be enrolled in elementary or secondary school, no previous training in Basic Life Support (BLS), and signing the informed consent and assent forms. Exclusion criteria will be participants who have already had CPR training before and those who cannot attend all planned activities. CPR is not currently part of the Brazilian educational curriculum in elementary and high school institutions.The training was developed following a pattern that included: welcoming the children, obtaining demographic data (weight, height, bicep circumference, palmar strength test), qualitative evaluation of the student's expectations in a written way, evaluation of the theoretical knowledge pre-test through a Serious Game(SGT0) developed by the researchers and published previously contemplating five elements (recognition of unconsciousness, call for help, initiate fast and strong chest compressions, maintain compressions at least 100 to 120 per minute, DEA), video-based training, post-test Serious Game(SGT1), post-course written qualitative perception and evaluation for 1 minute with QCPR manikin. All participants will receive 60 minutes video-based training CPR, practicing while watching based on American Heart Association (AHA) CPR in Schools Training Kit™ and 10 minutes training with continuous chest compressions (CCC) with audio feedback. The training sessions were conducted with classes of 20 participants during the school period. Mini Little Anne Manikin (Laerdal, Norway) and Little Anne QCPR® (Laerdal Medical Inc., Stavanger, Norway) with real-time feedback software (QCPR training 4.13.3, Laerdal Medical Inc., Stavanger, Norway) were used for training. Certified Basic Life Support instructors (AHA) conducted the training based on 2020 resuscitation guidelines with a ratio of 10:1 schoolchild to instructors.Categorical variables are presented as absolute and relative frequencies. Continuous variables are presented as median with interquartile range (IQR). Comparisons will be made between the groups: group 1 (age between 7 to 10 years) versus group 2 (age between 11 to 17 years), public versus private school, female sex versus male, and QCPR score <70 versus 70. Categorical variables were compared with chi-square test or Fisher exact test when appropriate. Continuous variables were compared using independent t test or Mann-Whitney U test in case of non-normal distribution. Normality was assessed by the Kolmogorov-Smirnov test. Two-tailed tests were used, and when p <0.05, the test was considered statistically significant. All analyses were conducted using R software version 4.1.0 (R Foundation for Statistical Computing).

ELIGIBILITY:
* a scientific cooperation agreement with university,
* being enrolled in elementary or secondary school
* no previous training in Basic Life Support (BLS)

Exclusion Criteria:

* no sign informed consent and assent.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — 7 to17 years old
Enrollment: 336 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Depth compression | one hour after training
  variability in compression depth among different age groups, taking into account physical attributes in millimetres

SECONDARY OUTCOMES:
Knowledge serious game | one hour after training
  difference between game score before and after training CPR (minimum 0 to maximun 500)

CONTACTS AND LOCATIONS:
Locations (1):
- Uri Adrian Prync Flato, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No